CLINICAL TRIAL: NCT03098199
Title: AMH and Dosing Regimens for Initial IVF Stimulation Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Specialists of New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 597102-3
Record Dates: First submitted 2017-03-01; First posted 2017-03-31 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Infertility
Keywords: Antimullerian Hormone; In vitro fertilization; Medications; Dosing
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Follicle Stimulating Hormone; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AMH<1.5, 300IU Gonal-F + 150 IU Menopur (Experimental): dosage at 300IU Gonal-F + 150IU Menopur
  Interventions: Drug: 300IU Gonal-F; Drug: 150IU Menopur
- AMH 1.6-2.5, 225IU Gonal-F+75IU Menopur (Experimental): dosage of 225IU Gonal-F + 75IU Menopur
  Interventions: Drug: 225IU Gonal-F; Drug: 75IU Menopur
- AMH 2.6-6.9, 150IU Gonal-F+75IU Menopur (Experimental): start dosage of 150IU Gonal-F and 75IU Menopur
  Interventions: Drug: 75IU Menopur; Drug: 150IU Gonal-F
- AMH >=7.0, 75IU Gonal-F+75U Menopur (Experimental): start dosage of 75IU Gonal-F and 75U Menopur
  Interventions: Drug: 75IU Menopur; Drug: 75IU Gonal-F

INTERVENTIONS:
Drug: 300IU Gonal-F — <1.5 AMH group
  Other Names: follitropin
  Arms: AMH<1.5, 300IU Gonal-F + 150 IU Menopur
Drug: 150IU Menopur — <1.5 AMH group
  Other Names: menotropin
  Arms: AMH<1.5, 300IU Gonal-F + 150 IU Menopur
Drug: 225IU Gonal-F — 1.6-2.5 AMH group
  Arms: AMH 1.6-2.5, 225IU Gonal-F+75IU Menopur
Drug: 75IU Menopur — 1.6-2.5 AMH group 2.6-6.9 AMH group >7.0 AMH group
  Arms: AMH 1.6-2.5, 225IU Gonal-F+75IU Menopur; AMH 2.6-6.9, 150IU Gonal-F+75IU Menopur; AMH >=7.0, 75IU Gonal-F+75U Menopur
Drug: 150IU Gonal-F — 2.6-6.9 AMH group
  Arms: AMH 2.6-6.9, 150IU Gonal-F+75IU Menopur
Drug: 75IU Gonal-F — >7.0 AMH group
  Arms: AMH >=7.0, 75IU Gonal-F+75U Menopur

SUMMARY:
This is a research study on a hormone in women called anti-mullerian hormone (AMH) an indicator of the amount of egg reserve in the ovaries. The research involves a blood draw to determine the AMH level. This knowledge will help the investigators decide a dosage of gonadotropins, the hormones used to stimulate the production of more than one egg for use in an in vitro fertilization (IVF) cycle. The amount of gonadotropin given has to be tailored to each individual participant. The investigators can use information about the participant and the hormone levels to determine this dosage and the chances of becoming pregnant as a result of IVF treatment. The reason the investigators are doing this research is to find out if basing the gonadotropin dosage solely on the participant's AMH level will give the investigators a better result than the previous method based on age and other hormone levels.

DETAILED DESCRIPTION:
Background / Rationale Anti-Müllerian Hormone (AMH) has been established as a valuable biomarker of ovarian reserve. It is a glycoprotein produced by granulosa cells of the ovary; it regulates the development of the primary follicle while inhibiting further recruitment of other surrounding follicles. Day 3 FSH and basal antral follicle count have traditionally been used to assess ovarian reserve and while they remain excellent predictors of poor ovarian response, they have not been shown to predict IVF success rates. Given the association between AMH and ovarian reserve, it has been proposed that AMH level can be used to predict ovarian response to gonadotropin stimulation and also, IVF success rates. An inverse relationship between AMH and total gonadotropin dosage has previously been demonstrated. As such, the concept of tailoring stimulation protocols to the patient's potential for oocyte production based on AMH level has gained favor. Individualization allows the practitioner to use the minimum dosage of medication required for maximum response, while limiting the risk of ovarian hyperstimulation syndrome. The question becomes how to determine the dosage of medication required for each AMH level and what effect will this have on clinical outcomes?

Hypothesis 1) Knowledge of AMH level used to determine medication dosage at the start of the stimulation cycle will result in a higher oocyte yield at the time of retrieval, higher clinical pregnancy rate, and higher live birth rate.

2) Knowledge of AMH level used to determine initial medication dosage at the start of the stimulation cycle will result in a fewer number of dosage changes mid-cycle.

3) Knowledge of AMH level prior to the start of a stimulation cycle will result in the use of a different initial stimulation dose compared to cycles in which the AMH is unknown.

4) Knowledge of AMH level used to determine medication dosage prior to the start of the stimulation cycle will result in a lower rate of ovarian hyperstimulation syndrome (OHSS). (Defined as >=20 oocytes/follicles) 5) Knowledge of AMH level used to determine medication dosage prior to the start of the stimulation cycle will result in a lower rate of cancelled cycles.

Methods and Procedures. The AMH level for all patients will be assessed at the initial fertility evaluation for each patient.

Patients will undergo controlled ovarian hyperstimulation (COH) with a GnRH antagonist protocol. They will begin COH on day 3 of their menstrual cycle or they may need to begin with approximately one week of oral contraceptives. After one week, the patients will stop taking oral contraceptives if their ovaries appear quiescent on transvaginal ultrasound and their serum E2 levels are low. These patients will then begin COH three days later. Gonadotropin dosage will be determined at the start of the cycle by AMH level.

Dosages will be adjusted, beginning on the third day of gonadotropins, based on clinical response, determined by serum hormone levels and transvaginal ultrasound of the ovaries throughout the cycle. The patient will begin taking the GnRH antagonist, Ganirelix or Cetrotide, when the lead follicle measures ≥14mm on transvaginal ultrasound. Patients will be triggered with Lupron, hCG, or both when the lead follicle measures ≥20mm on transvaginal ultrasound. All medications are administered via subcutaneous injections.

Transvaginal ultrasound-guided oocyte retrieval will be performed 36 hours after the trigger medication(s) is administered. Cycles with a poor ovarian response, defined as <3 follicles and/or a peak estradiol level <600 pg/mL, will be canceled.

Patients will undergo culture day 5 embryo transfer; number of embryos transferred will be according to ASRM guidelines. If the patient exhibits symptoms of OHSS, she will discontinue luteal phase support and will not have an embryo transfer, and all good quality blastocyst mbryos will be cryopreserved. All patients eligible for embryo transfer will continue the luteal phase support protocol until the serum hCG pregnancy test 14 days post-retrieval. If the serum hCG is <5 mIU/mL, luteal phase support will be discontinued. If the serum hCG is ≥5 mIU/mL, Estrace will continue to be taken until 8 weeks gestation and Endometrin or intramuscular progesterone in oil will continue to be used until 10 weeks gestation. At this point, patient is released to the care of the obstetrician. The patient or the obstetrician will be contacted for pregnancy outcome data.

ELIGIBILITY:
Inclusion Criteria:

* first cycle of IVF with transfer of fresh embryo

Exclusion Criteria:

* use of non-autologous oocytes; prior diagnosis of premature ovarian failure or diminished ovarian reserve; BMI>= 40; cryopreservation cycles; smokers; use of PGS/PGD; use of surgically retrieved sperm or patients with severe male factor; and oocyte- or embryo-banking cycles

Ages: 25 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | two years
  Clinical pregnancy rate is defined as the number of pregnancies with the presence of an intrauterine gestational sac seen on transvaginal ultrasound by six weeks gestation divided by the number of completed embryo transfers.

SECONDARY OUTCOMES:
Oocyte yield | two years
  number of follicles produced

CONTACTS AND LOCATIONS:
Overall Officials: Linda Sung, MD, Principal Investigator — Reproductive Specialists of New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anderson RA, Nelson SM, Wallace WH. Measuring anti-Mullerian hormone for the assessment of ovarian reserve: when and for whom is it indicated? Maturitas. 2012 Jan;71(1):28-33. doi: 10.1016/j.maturitas.2011.11.008. Epub 2011 Nov 26. PMID 22119275
- [Background] de Vet A, Laven JS, de Jong FH, Themmen AP, Fauser BC. Antimullerian hormone serum levels: a putative marker for ovarian aging. Fertil Steril. 2002 Feb;77(2):357-62. doi: 10.1016/s0015-0282(01)02993-4. PMID 11821097
- [Background] Freour T, Mirallie S, Colombel A, Bach-Ngohou K, Masson D, Barriere P. Anti-mullerian hormone: clinical relevance in assisted reproductive therapy. Ann Endocrinol (Paris). 2006 Dec;67(6):567-74. doi: 10.1016/s0003-4266(06)73008-6. PMID 17194966
- [Background] Gleicher N, Kim A, Weghofer A, Barad DH. Toward a better understanding of functional ovarian reserve: AMH (AMHo) and FSH (FSHo) hormone ratios per retrieved oocyte. J Clin Endocrinol Metab. 2012 Mar;97(3):995-1004. doi: 10.1210/jc.2011-2403. Epub 2011 Dec 14. PMID 22170712
- [Background] Jayaprakasan K, Campbell B, Hopkisson J, Johnson I, Raine-Fenning N. A prospective, comparative analysis of anti-Mullerian hormone, inhibin-B, and three-dimensional ultrasound determinants of ovarian reserve in the prediction of poor response to controlled ovarian stimulation. Fertil Steril. 2010 Feb;93(3):855-64. doi: 10.1016/j.fertnstert.2008.10.042. Epub 2008 Nov 30. PMID 19046583
- [Background] Kwee J, Schats R, McDonnell J, Themmen A, de Jong F, Lambalk C. Evaluation of anti-Mullerian hormone as a test for the prediction of ovarian reserve. Fertil Steril. 2008 Sep;90(3):737-43. doi: 10.1016/j.fertnstert.2007.07.1293. Epub 2007 Oct 17. PMID 17923131
- [Background] Panchal S, Nagori C. Comparison of anti-mullerian hormone and antral follicle count for assessment of ovarian reserve. J Hum Reprod Sci. 2012 Sep;5(3):274-8. doi: 10.4103/0974-1208.106340. PMID 23531919
- [Background] Tremellen KP, Kolo M, Gilmore A, Lekamge DN. Anti-mullerian hormone as a marker of ovarian reserve. Aust N Z J Obstet Gynaecol. 2005 Feb;45(1):20-4. doi: 10.1111/j.1479-828X.2005.00332.x. PMID 15730360
- [Background] van Rooij IA, Broekmans FJ, te Velde ER, Fauser BC, Bancsi LF, de Jong FH, Themmen AP. Serum anti-Mullerian hormone levels: a novel measure of ovarian reserve. Hum Reprod. 2002 Dec;17(12):3065-71. doi: 10.1093/humrep/17.12.3065. PMID 12456604
- [Background] Biasoni V, Patriarca A, Dalmasso P, Bertagna A, Manieri C, Benedetto C, Revelli A. Ovarian sensitivity index is strongly related to circulating AMH and may be used to predict ovarian response to exogenous gonadotropins in IVF. Reprod Biol Endocrinol. 2011 Aug 9;9:112. doi: 10.1186/1477-7827-9-112. PMID 21824441
- [Background] Choi MH, Yoo JH, Kim HO, Cha SH, Park CW, Yang KM, Song IO, Koong MK, Kang IS. Serum anti-Mullerian hormone levels as a predictor of the ovarian response and IVF outcomes. Clin Exp Reprod Med. 2011 Sep;38(3):153-8. doi: 10.5653/cerm.2011.38.3.153. Epub 2011 Sep 30. PMID 22384435
- [Background] Elgindy EA, El-Haieg DO, El-Sebaey A. Anti-Mullerian hormone: correlation of early follicular, ovulatory and midluteal levels with ovarian response and cycle outcome in intracytoplasmic sperm injection patients. Fertil Steril. 2008 Jun;89(6):1670-6. doi: 10.1016/j.fertnstert.2007.05.040. Epub 2007 Jul 20. PMID 17658520
- [Background] Honnma H, Baba T, Sasaki M, Hashiba Y, Oguri H, Fukunaga T, Endo T, Asada Y. Different ovarian response by age in an anti-Mullerian hormone-matched group undergoing in vitro fertilization. J Assist Reprod Genet. 2012 Feb;29(2):117-25. doi: 10.1007/s10815-011-9675-9. Epub 2011 Nov 16. PMID 22086616
- [Background] La Marca A, Giulini S, Tirelli A, Bertucci E, Marsella T, Xella S, Volpe A. Anti-Mullerian hormone measurement on any day of the menstrual cycle strongly predicts ovarian response in assisted reproductive technology. Hum Reprod. 2007 Mar;22(3):766-71. doi: 10.1093/humrep/del421. Epub 2006 Oct 27. PMID 17071823
- [Background] Muttukrishna S, McGarrigle H, Wakim R, Khadum I, Ranieri DM, Serhal P. Antral follicle count, anti-mullerian hormone and inhibin B: predictors of ovarian response in assisted reproductive technology? BJOG. 2005 Oct;112(10):1384-90. doi: 10.1111/j.1471-0528.2005.00670.x. PMID 16167941
- [Background] Nardo LG, Gelbaya TA, Wilkinson H, Roberts SA, Yates A, Pemberton P, Laing I. Circulating basal anti-Mullerian hormone levels as predictor of ovarian response in women undergoing ovarian stimulation for in vitro fertilization. Fertil Steril. 2009 Nov;92(5):1586-93. doi: 10.1016/j.fertnstert.2008.08.127. Epub 2008 Oct 18. PMID 18930213
- [Background] Singh N, Malik E, Banerjee A, Chosdol K, Sreenivas V, Mittal S. "Anti-Mullerian Hormone: Marker for Ovarian Response in Controlled Ovarian Stimulation for IVF Patients": A First Pilot Study in the Indian Population. J Obstet Gynaecol India. 2013 Aug;63(4):268-72. doi: 10.1007/s13224-012-0318-6. Epub 2013 Feb 22. PMID 24431654
- [Background] Wu CH, Chen YC, Wu HH, Yang JG, Chang YJ, Tsai HD. Serum anti-Mullerian hormone predicts ovarian response and cycle outcome in IVF patients. J Assist Reprod Genet. 2009 Jul;26(7):383-9. doi: 10.1007/s10815-009-9332-8. PMID 19768530
- [Background] Alviggi C, Humaidan P, Ezcurra D. Hormonal, functional and genetic biomarkers in controlled ovarian stimulation: tools for matching patients and protocols. Reprod Biol Endocrinol. 2012 Feb 6;10:9. doi: 10.1186/1477-7827-10-9. PMID 22309877
- [Background] Bosch E, Ezcurra D. Individualised controlled ovarian stimulation (iCOS): maximising success rates for assisted reproductive technology patients. Reprod Biol Endocrinol. 2011 Jun 21;9:82. doi: 10.1186/1477-7827-9-82. PMID 21693025
- [Background] Broer SL, Dolleman M, Opmeer BC, Fauser BC, Mol BW, Broekmans FJ. AMH and AFC as predictors of excessive response in controlled ovarian hyperstimulation: a meta-analysis. Hum Reprod Update. 2011 Jan-Feb;17(1):46-54. doi: 10.1093/humupd/dmq034. Epub 2010 Jul 28. PMID 20667894
- [Background] Fleming R, Broekmans F, Calhaz-Jorge C, Dracea L, Alexander H, Nyboe Andersen A, Blockeel C, Jenkins J, Lunenfeld B, Platteau P, Smitz J, de Ziegler D. Can anti-Mullerian hormone concentrations be used to determine gonadotrophin dose and treatment protocol for ovarian stimulation? Reprod Biomed Online. 2013 May;26(5):431-9. doi: 10.1016/j.rbmo.2012.02.027. Epub 2013 Feb 4. PMID 23507133
- [Background] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Background] Martinez F, Clua E, Carreras O, Tur R, Rodriguez I, Barri PN. Is AMH useful to reduce low ovarian response to GnRH antagonist protocol in oocyte donors? Gynecol Endocrinol. 2013 Aug;29(8):754-7. doi: 10.3109/09513590.2013.801443. Epub 2013 Jun 12. PMID 23758138
- [Background] Nakhuda GS, Douglas NC, Thornton MH, Guarnaccia MM, Lobo R, Sauer MV. Anti-Mullerian hormone testing is useful for individualization of stimulation protocols in oocyte donors. Reprod Biomed Online. 2010 Jan;20(1):42-7. doi: 10.1016/j.rbmo.2009.10.009. Epub 2009 Oct 30. PMID 20158986
- [Background] Nelson SM, Yates RW, Fleming R. Serum anti-Mullerian hormone and FSH: prediction of live birth and extremes of response in stimulated cycles--implications for individualization of therapy. Hum Reprod. 2007 Sep;22(9):2414-21. doi: 10.1093/humrep/dem204. Epub 2007 Jul 18. PMID 17636277
- [Background] Yates AP, Rustamov O, Roberts SA, Lim HY, Pemberton PW, Smith A, Nardo LG. Anti-Mullerian hormone-tailored stimulation protocols improve outcomes whilst reducing adverse effects and costs of IVF. Hum Reprod. 2011 Sep;26(9):2353-62. doi: 10.1093/humrep/der182. Epub 2011 Jun 13. PMID 21672928